CLINICAL TRIAL: NCT03172507
Title: Phenotypic and Epigenetic "Trained Immunity" Characteristics of Hematopoietic Stem and Progenitor Cells in Patients With Established Atherosclerosis
Brief Title: The Role of Stem Cells on Immune Cells in the Development of Cardiovascular Diseases
Acronym: ATHEROSTEM
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL58806.091.16
Record Dates: First submitted 2017-03-31; First posted 2017-06-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-10

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Hematopoietic Stem Cells
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma and bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Atherosclerosis group: Patients with significant coronary artery disease.
- Control group: Healthy controls without confirmed coronary artery disease.

SUMMARY:
An observational pilot proof-of-principle study. 15 patients with significant coronary artery disease and 15 matched controls. To investigate whether long-term activation of the innate immune system, named 'trained innate immunity', occurs at the level of the bone marrow progenitor cells in patients with significant coronary artery disease and whether this correlates with the proinflammatory phenotype of monocytes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years
* With or without significant coronary artery disease on CCTA
* Written informed consent

Exclusion Criteria:

* Chronic infections
* Diabetes mellitus
* Medical history of any disease associated with immune deficiency
* Clinically significant infections within 3 months prior to study entry
* Recent hospital admission or surgery with general anaesthesia
* Known chronic kidney or liver disease
* Previous vaccination within 3 months prior to study entry
* Inability to personally provide written informed consent
* Inability to undergo PET-CT scanning
* Chronic use of anti-inflammatory drugs such as NSAIDs
* History of haematological malignant disease
* Documented bleeding diathesis or thrombocytopenia
* Pregnancy

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 15 patients with significant coronary artery disease and 15 patients without significant coronary artery disease. Patients who have been presented to the cardiology departments of the CWZ hospital or Radboud University Medical Centre and have undergone CCTA in the past two years are eligible to participate if they meet the in- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Phenotypical characteristics of HSPC's | Study day 2 for patients
  Phenotypical characteristics of HSPC's populations of patients with and without significant coronary artery disease by flowcytometry in percentages.
Cytokine response of circulating monocytes | Study day 2 for patients
  Cytokine response of monocytes of patients with and without significant coronary artery disease after 24 hour stimulation with several stimuli measured in cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Niels P. Riksen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Department of cardiology, CWZ, Nijmegen, Gelderland
  - Department of cardiology, Radboudumc, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noz MP, Bekkering S, Groh L, Nielen TM, Lamfers EJ, Schlitzer A, El Messaoudi S, van Royen N, Huys EH, Preijers FW, Smeets EM, Aarntzen EH, Zhang B, Li Y, Bremmers ME, van der Velden WJ, Dolstra H, Joosten LA, Gomes ME, Netea MG, Riksen NP. Reprogramming of bone marrow myeloid progenitor cells in patients with severe coronary artery disease. Elife. 2020 Nov 10;9:e60939. doi: 10.7554/eLife.60939. PMID 33168134